CLINICAL TRIAL: NCT00387920
Title: A Phase I Study of Sunitinib (SU11248), an Oral Multi-Targeted Tyrosine Kinase Inhibitor, in Children With Refractory Solid Tumors
Brief Title: Sunitinib in Treating Young Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00361; NCI-2009-00361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000507414; COG-ADVL0612; NCI-07-C-0220; ADVL0612 (Other: COG Phase I Consortium); ADVL0612 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Central Nervous System Metastases; Childhood Central Nervous System Choriocarcinoma; Childhood Central Nervous System Embryonal Tumor; Childhood Central Nervous System Germ Cell Tumor; Childhood Central Nervous System Germinoma; Childhood Central Nervous System Mixed Germ Cell Tumor; Childhood Central Nervous System Teratoma; Childhood Central Nervous System Yolk Sac Tumor; Recurrent Childhood Central Nervous System Embryonal Tumor; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — Sunitinib

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): PART A: Patients receive oral sunitinib malate once daily on days 1-28 days. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  PART B: Patients receive sunitinib malate capsule contents sprinkled over applesauce or yogurt once daily on days 1-28. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. After the first course, patients may switch to capsule formulation for convenience.
  Interventions: Drug: sunitinib malate; Other: pharmacological study; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Undergo DCE-MRI
  Other Names: DCE-MRI
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of sunitinib in treating young patients with refractory solid tumors. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and recommended phase II dose of sunitinib malate in pediatric patients with refractory solid tumors.

II. Determine the toxicity of this regimen in these patients. III. Characterize the pharmacokinetics of this regimen in these patients. IV. Evaluate the tolerability and pharmacokinetic profile of sunitinib malate capsule contents sprinkled over applesauce or yogurt using the recommended phase II dose.

SECONDARY OBJECTIVES:

I. Determine, preliminarily, the antitumor effects of this regimen in these patients.

II. Describe changes in peripheral blood monocyte counts, circulating endothelial cells, and plasma angiogenic factors during treatment with sunitinib malate.

III. Explore changes in tumor vascular permeability using dynamic contrast-enhanced (DCE)-magnetic resonance imaging (MRI) in patients receiving sunitinib malate.

OUTLINE: This is a multicenter, dose-escalation study (part A) followed by a pediatric-friendly formulation study (part B).

PART A: Patients receive oral sunitinib malate once daily on days 1-28 days. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of sunitinib malate until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PART B: Patients receive sunitinib malate capsule contents sprinkled over applesauce or yogurt once daily on days 1-28. Treatment repeats every 42 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. After the first course, patients may switch to capsule formulation for convenience.

NOTE: Patients will not receive sunitinib malate on day 2 of the first course to allow for pharmacokinetic testing.

Blood is collected on days 1, 7, 14, 21, and 28 of course 1 for pharmacokinetic studies using liquid chromatography/mass spectrometry.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor (not required for patients with intrinsic brain stem tumors or optic pathway gliomas)

  * Recurrent or refractory disease
* Measurable or evaluable disease
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life exists
* Patients with metastatic bone marrow disease are eligible but are not evaluable for hematologic toxicity

  * Must not be refractory to red blood cell or platelet transfusions
* Primary CNS tumors or known CNS metastases allowed

  * Neurological deficits must have been relatively stable for ≥ 1 week before study enrollment
  * No imaging evidence of prior intracranial hemorrhage
  * No evidence of new CNS hemorrhage on baseline MRI obtained within 14 days before study enrollment (ECHO gradient MRI sequences per institutional guidelines required for evaluation of CNS hemorrhage)

    * The presence of small punctuate CNS hemorrhage on these scans will exclude a patient from participation
* No known bone marrow metastatic disease
* No tumors involving the pleural surface
* Karnofsky performance status (PS) 50-100% (> 10 years of age) OR Lansky PS 50-100% (≤ 10 years of age)
* Absolute neutrophil count ≥ 1,000/mm³*
* Platelet count ≥ 100,000/mm³ (transfusion independent)*
* Hemoglobin ≥ 8.0 g/dL (transfusions allowed)*
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine based on age/gender as follows:

  * No greater than 0.8 mg/dL (2 to 5 years of age)
  * No greater than 1 mg/dL (6 to 9 years of age)
  * No greater than 1.2 mg/dL (10 to 12 years of age)
  * No greater than 1.5 mg/dL (male) OR 1.4 mg/dL (female) (13 to 15 years of age)
  * No greater than 1.7 mg/dL (male) OR 1.4 mg/dL (female) (≥ 16 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for liver metastases)
* Albumin ≥ 2 g/dL
* LVEF or shortening fraction normal
* Corrected QT interval ≤ 450 msec
* Amylase ≤ 1.5 times ULN
* Lipase ≤ 1.5 times ULN
* Body surface area ≥ 0.5 m² (≥ 0.4 m² for part B)
* Blood pressure within ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled infection
* Able to swallow sunitinib malate capsules (part A only)
* No pre-existing thyroid abnormality (hyper- or hypothyroidism) with unstable thyroid function
* No prior CNS hemorrhage
* No history of allergic reaction attributed to sunitinib malate or component of sunitinib malate capsules
* No allergy to both applesauce and yogurt (part B only)
* Recovered from prior therapy
* No prior sunitinib malate
* No prior anthracycline (any dose)
* No prior radiotherapy to a radiation field that included the heart(including total body or craniospinal irradiation)
* At least 3 months since prior stem cell transplantation or rescue (without total-body irradiation) and no evidence of graft-vs-host disease
* At least 2 weeks since prior local, palliative, small-port radiotherapy (at least 6 months for radiation to ≥ 50% of pelvis)
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 3 weeks since prior myelosuppressive therapy (6 weeks for nitrosoureas)
* At least 1 week since prior antineoplastic biologic agents
* At least 1 week since prior and no concurrent hematopoietic growth factors
* At least 12 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Hypericum perforatum (St. John's wort)
  * Efavirenz
  * Tipranavir
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Azole antifungals (e.g., itraconazole or ketoconazole)
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * HIV protease inhibitors (e.g., indinavir, saquinavir, ritonavir, atazanavir, or nelfinavir)
  * Delavirdine
* No more than 1 concurrent antihypertensive agent
* No concurrent major surgery
* No concurrent antithrombotic or antiplatelet agents, including any of the following:

  * Warfarin
  * Heparin
  * Low molecular weight heparin
  * Acetylsalicylic acid (aspirin)
  * Ibuprofen
  * Other nonsteroidal anti-inflammatory drugs
* No concurrent medication for the treatment of hypertension
* No other concurrent investigational drugs
* No other concurrent anticancer agents, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2006-10; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
MTD and recommended phase II dose | During course 1 of therapy
  MTD will be the maximum dose at which fewer than one-third of patients experience dose-limiting toxicity (DLT).
Adverse events as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Weekly during course 1, assessed up to 35 days
Pharmacokinetics of sunitinib malate using liquid spectrometry/mass spectroscopy methods | At baseline and days 1, 7, 14, 21, and 28 of course 1
Tolerability and pharmacokinetic profile of capsule contents sprinkled over applesauce or yogurt | At baseline and days 1, 7, 14, 21, and 28 of course 1

SECONDARY OUTCOMES:
Correlative studies | Days 1 and 28 of course 1
  The laboratory, radiology, and pathology correlative studies are largely expected to be exploratory. Mean and median values will be reported at each time point for circulating endothelial cells, monocyte count, plasma angiogenic markers, and DCE-MRI vascular permeability. Depending on the distribution of data, either the paired t-test or Wilcoxon signed rank test will be used to evaluate for statistically significant changes in these markers from pre-treatment to post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, Principal Investigator — COG Phase I Consortium
Locations (17):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Childrens Hospital of Orange County, Orange, California
  - UCSF-Mount Zion, San Francisco, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Wang E, DuBois SG, Wetmore C, Verschuur AC, Khosravan R. Population Pharmacokinetics of Sunitinib and its Active Metabolite SU012662 in Pediatric Patients with Gastrointestinal Stromal Tumors or Other Solid Tumors. Eur J Drug Metab Pharmacokinet. 2021 May;46(3):343-352. doi: 10.1007/s13318-021-00671-7. Epub 2021 Apr 14. PMID 33852135
- [Derived] Wang E, DuBois SG, Wetmore C, Khosravan R. Population pharmacokinetics-pharmacodynamics of sunitinib in pediatric patients with solid tumors. Cancer Chemother Pharmacol. 2020 Aug;86(2):181-192. doi: 10.1007/s00280-020-04106-z. Epub 2020 Jul 4. PMID 32623479